CLINICAL TRIAL: NCT05517681
Title: Application of ICG in Lymph Node Dissection During Radical Resection of Rectal Cancer With Preserved Autonomic Nerves Around LCA and IMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Qinhuangdao (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20210130
Record Dates: First submitted 2022-08-23; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Indocyanine Green
Keywords: Indocyanine Green; Rectal Cancer; Autonomic nerve; Inferior mesenteric artery; Left colic artery; lymph nodes
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-ICG Group (Placebo Comparator): Laparoscopic radical resection of rectal cancer was performed routinely without ICG injection
  Interventions: Other: non-ICG
- ICG Group (Experimental): ICG was injected preoperatively via anoscope or anal dilator in the mucosal layer around the tumor, and surgical treatment was performed after visualization. The surgical approach was performed by laparoscopic radical rectal cancer with an intermediate approach step.The IMA root is treated with low ligation of the IMA, while lymph node dissection is performed while preserving the autonomic nerves around the IMA
  Interventions: Drug: ICG

INTERVENTIONS:
Other: non-ICG — Laparoscopic radical resection of rectal cancer was performed routinely without ICG injection. The separation should extend from the center to the left, reaching the left paracolic sulcus lateral to the genital vessels. The Superior hypogastric nerve is protected by freeing it at the angle of the common iliac artery on both sides, afterwards, the vessel is free along the surface of the plexus from caudal to cephalic side to reach the root of the IMA. Switching lymph node visualization patterns. Based on the operator's experience and the extent of lymph node visualization, the lymph nodes at the root of the IMA were removed with an ultrasonic knife . The dissection continues caudally along the IMA, preserving the arterial sheath. Expose the left colonic artery, superior rectal artery, and sigmoid artery, maximum preservation of the IMA peripheral plexus while clearing their surrounding lymph nodes.
  Arms: non-ICG Group
Drug: ICG — Dilute ICG to 2.5 mg/ml with its accompanying sterilized water for injection. Slow injection with a 1ml syringe in 4 parts of the tumor，Inject 0.25ml per site . Procedure started after lymph node visualization.The operation was consistent with the control group.
  Arms: ICG Group

SUMMARY:
Indocyanine green NIR imaging is valuable for lymph node dissection in D3 radical surgery for rectal cancer. It can guide the intraoperative improvement of lymph node dissection based on the preservation of LCA and peripheral autonomic nerves of IMA. This not only reduces the occurrence of postoperative complications and promotes rapid postoperative recovery, but also provides a more precise and individualized comprehensive treatment plan for patients after surgery. In addition，this trial also demonstrated that ICG is safe and feasible for use in rectal cancer

DETAILED DESCRIPTION:
The pathological data of 96 patients with rectal cancer from September 2020 - July 2022 were collected from the First Hospital of Qinhuangdao City.In 51 of these patients, ICG was injected preoperatively via anoscope or anal dilator in the mucosal layer around the tumor, and surgical treatment was performed after visualization. The surgical approach was performed by laparoscopic radical rectal cancer with an intermediate approach step.The IMA root is treated with low ligation of the IMA, while lymph node dissection is performed while preserving the autonomic nerves around the IMA. The other 45 patients were not injected with ICG, and the procedure was performed as before.The occurrence of postoperative complications was recorded, and the detection of lymph nodes was also compared between the two groups, as well as the intraoperative situation and postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

1. The preoperative colonoscopic pathological diagnosis was clearly rectal cancer and no malignant tumor in other sites.
2. Good preoperative general condition, no serious cardiopulmonary, hepatic, renal or other major comorbidities before surgery
3. Radical rectal cancer surgery with preservation of LCA and peripheral autonomic nerves of IMA in patients
4. No contraindications to surgery
5. No history of ICG or iodide allergy

Exclusion Criteria:

-

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
The number of cleared IMA root lymph nodes | immediately after surgery
  A group of lymph nodes surrounding the inferior mesenteric artery between the origin of the artery and the left colic artery
The total number of cleared lymph nodes | immediately after surgery
  The sum of IMA root lymph nodes and lymph nodes surrounding the tumor area
The number of positive lymph nodes | immediately after surgery
  There are metastatic tumor cells in the lymph nodes

SECONDARY OUTCOMES:
Quality of postoperative recovery | Up to 7 days after surgery
  days of postoperative hospitalization, days of retention of the urinary catheter, days of retention of abdominal drainage tube, time of first fluid intake and IPSS score
The incidence of postoperative complications | Up to 7 days after surgery
  mild or severe urogenital disorders, anastomotic leakage, anastomotic bleeding, abdominal infection, intestinal obstruction.

CONTACTS AND LOCATIONS:
Overall Officials: liuhanchong Hanchong Liu, Study Chair — The First Hospital of Qinhuangdao
Locations (1):
- The First hosptial of Qinhuangdao, Qinhuangdao, China

IPD SHARING:
Plan to Share IPD: No